CLINICAL TRIAL: NCT02971540
Title: Comparative, Randomized Trial of SPI-directed Intravenous Analgesia Using Metamizole With Tramadol Versus Preemptive Wound Infiltration Using 0,2 % Ropivacaine With Fentanyl or 0,2 % Bupivacaine With Fentanyl for Lumbar Discectomy
Brief Title: SPI-directed Analgesia for Lumbar Discectomy
Acronym: SPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Michał Stasiowski, Principal Investigator, 2Department of Anaesthesiology and Intensive Therapy, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SilesianMUKOAiIT1
Record Dates: First submitted 2016-11-02; First posted 2016-11-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Lumbar Disc Disease
Keywords: Surgical Pleth Index (SPI); General Anaesthesia (GA),; Numerical Rating Scale (NRS); Adequacy of Anaesthesia (AoA; Spectral Entropy (SE); Local Anesthetic (LA)
MeSH Terms: conditions — Intervertebral disc disease; Early-onset ataxia with oculomotor apraxia and hypoalbuminemia | interventions — Dipyrone; Tramadol; Bupivacaine; Ropivacaine; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- bupivacaine, LA, solution (Experimental): an a local anesthetic administered for local wound infiltration on each side in a single dose of 10 ml of 0,2% solution per segment of vertrebral columne with potential duration time of up to 8 hours according to manufacturers data
  Interventions: Drug: Metamizol; Drug: Tramadol; Drug: Ropivacaine; Other: control group
- ropivacaine, LA, solution (Experimental): an a local anesthetic administered for local wound infiltration on each side in a single dose of 10 ml of 0,2% solution per segment of vertrebral columne with potential duration time of up to 8 hours according to manufacturers data
  Interventions: Drug: Metamizol; Drug: Tramadol; Drug: Bupivacaine; Other: control group
- metamizol, analgesic, solution (Experimental): an analgesic drug administered intravenously for pre-emptive analgesia in a initial dose of 1-1,25g with potential duration time of up to 6 hours according to manufacturers data
  Interventions: Drug: Bupivacaine; Drug: Ropivacaine; Other: control group
- tramadol, analgesic, solution (Experimental): a half-opioid drug administered intravenously for pre-emptive analgesia in a initial dose of 2 mg per kg of body weight with potential duration time of up to 6 hours according to manufacturers data
  Interventions: Drug: Metamizol; Drug: Tramadol; Drug: Bupivacaine; Drug: Ropivacaine
- control group (Experimental): no pre-emptive analgesia will be used.
  Interventions: Drug: Metamizol; Drug: Tramadol; Drug: Bupivacaine; Drug: Ropivacaine; Other: control group

INTERVENTIONS:
Drug: Metamizol — in group A patients will receive pre-emptive analgesia using intravenous infusion of metamizol in a single dose of 1-1,25 gram with following intravenous infusion of 5 grams per day.
  Other Names: Pyralgina
  Arms: bupivacaine, LA, solution; control group; ropivacaine, LA, solution; tramadol, analgesic, solution
Drug: Tramadol — in group A patients will receive pre-emptive analgesia using intravenous infusion of tramadol in a single dose of 2 mg per hg of body weight with following intravenous infusion of 400 mg per day.
  Other Names: Poltram
  Arms: bupivacaine, LA, solution; control group; ropivacaine, LA, solution; tramadol, analgesic, solution
Drug: Bupivacaine — patients in group BF will receive local wound infiltration with a solution of 0,2% bupivacaine in a volume of 10 ml per segment of vertrebral columne.
  Other Names: Bupiwakaina WZF
  Arms: control group; metamizol, analgesic, solution; ropivacaine, LA, solution; tramadol, analgesic, solution
Drug: Ropivacaine — patients in group RF will receive local wound infiltration with a solution of 0,2% ropivacaine in a volume of 10 ml per segment of vertrebral columne.
  Other Names: Ropimol
  Arms: bupivacaine, LA, solution; control group; metamizol, analgesic, solution; tramadol, analgesic, solution
Other: control group — patients will receive no pre-emptive analgesia. intraoperatively standard dose of fentanyl will be used.
  Arms: bupivacaine, LA, solution; control group; metamizol, analgesic, solution; ropivacaine, LA, solution

SUMMARY:
The aim of this randomized trial is to assess the efficacy of analgesia for lumbar discectomy and compare Numerical Rating Scale (NRS) with Surgical Pleth Index (SPI) for monitoring pain perception postoperatively.

Patients received either preemptive local tissue infiltration at surgical site using either 0,2% ropivacaine with fentanyl or 0,2% bupivacaine with fenthanyl or preemptive intravenous infusion using metamizole and tramadol.

DETAILED DESCRIPTION:
Monitoring depth of anaesthesia using spectral entropy (SE) and quality of neuromuscular block are routine in modern anaesthesia, whereas monitoring of analgesia still requires further studies. Recently, the Surgical Pleth Index (SPI) was added as a surrogate variable showing the nociception-antinociception balance into abovementioned parametres constituting a novel approach in monitoring patients intraoperatively, known as adequacy of anaesthesia (AoA) or tailor-made anaesthesia. This study aims at evaluating utility of SPI-directed analgesia in patients undergoing general anaesthesia (GA) where analgesia intraoperatively will be achieved either with regional preemptive wound infiltration using 0,2 % ropivacaine with fentanyl or 0,2 % bupivacaine with fentanyl or intravenous analgesia using continuous infusion of metamizole with tramadol for lumbar discectomy. Intraoperatively, SPI value will be recorded with sampling frequency of 1 minute. When SPI value reaches a level higher than 15 SPI points above basic level, a rescue dose of 1mg/kg body weight of fentanyl will be administered intravenously every 5 minutes until SPI value decreases to basic level calculated previously before operation started.

Additionally, the investigators will compare Numerical Rating Scale (NRS) with Surgical Pleth Index (SPI) values for monitoring the efficacy of analgesia postoperatively. After emergence from GA patients will be questioned in terms of their pain intensity in a scale 0-10. In the case of pain perception above 3, a bolus of 2mg of morphine will be administered intravenously every 10 minutes until pain perception will be lower than 4. SPI values will be recorded every 1 minute and analysed for aute pain (NRS 7-10), average (4-6) and mild pain perception intervals to assess if there exists a correlation between NRS and SPI.

In addition, some patients develop Failed Back Surgery Syndrome (FBSS) following lumbar surgeries so the investigators will aim to analyze if SPI-directed analgesia intra- and post-operatively reduces rate of FBSS. After 5 months after operation patient will be surveyed using melzack protocol to assess the rate of FBSS as well as symptoms of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study
* written consent to undergo general anaesthesia with local wound infiltration and surgery of discectomy

Exclusion Criteria:

* allergy to local anaesthetics
* necessity of administration of vasoactive drugs influencing SPI monitoring
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
pain perception intraoperatively | on-line based on SPI values
  The investigators will compare the efficacy of analgesia intraoperatively according to technique of analgesia used preoperatively: either local woung inflitration or intravenous infusion. The investigators will administer a resuce dose of fentanyl intravenously in a dose of 1 mcg per kg of body weight in the case when SPI value increases over 15 points in SPI scale every 5 minutes untill SPI value decreases back to baseline value

SECONDARY OUTCOMES:
pain perception postoperatively | 2 hours after discharge to postoperative unit.
  The investigators will compare the efficacy of analgesia postoperatively according to technique of analgesia used preoperatively: either local woung inflitration or intravenous infusion. The investigators use NRS and compare it with SPI values. Additionally, The investigators will observe SPI variations as a reaction to morphine administration intravenously in the case of acute or moderate pain.

OTHER OUTCOMES:
postoperative persistent pain | up to 6 months
  The investigators will compare the efficacy of analgesia postoperatively according to technique of analgesia used preoperatively: either local woung inflitration or intravenous infusion. The investigators will use melzack to assess the rate of the post-operative persistent pain. Patients will be invited to pay a control visit in the clinic and asked to describe their pain intensity and specify its characteristic using a set of adjectives characterizing their pain perception. Afterwards, pain perception of patients will be analyzed using specified scale when each adjective is attributed points and sum of points gathered in the questionaire indicates probability of presence of postoperative perception pain using melzack questionnaire.
postoperative FBSS | up to 6 months
  The investigators will compare the efficacy of analgesia postoperatively according to technique of analgesia used preoperatively: either local woung inflitration or intravenous infusion. The investigators will use FBSS scale to assess the presence of FBSS. Patients will be invited to pay a control visit in the clinic to be diagnosed for symptoms of FBSS: pain intensity, disability, depression scores, temperament and character profile determined by the visual analogue scale (VAS), Roland Morris Disability Index, Beck Depression Inventory, and Temperament and Character Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Michał J Stasiowski, M.D, Principal Investigator — Medical University of Silesia
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
article in AiIT in 2019,
Supporting Information: ICF

REFERENCES:
- [Background] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Background] Gruenewald M, Ilies C. Monitoring the nociception-anti-nociception balance. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):235-47. doi: 10.1016/j.bpa.2013.06.007. PMID 24012235
- [Background] Gruenewald M, Willms S, Broch O, Kott M, Steinfath M, Bein B. Sufentanil administration guided by surgical pleth index vs standard practice during sevoflurane anaesthesia: a randomized controlled pilot study. Br J Anaesth. 2014 May;112(5):898-905. doi: 10.1093/bja/aet485. Epub 2014 Feb 16. PMID 24535604
- [Background] Won YJ, Lim BG, Lee SH, Park S, Kim H, Lee IO, Kong MH. Comparison of relative oxycodone consumption in surgical pleth index-guided analgesia versus conventional analgesia during sevoflurane anesthesia: A randomized controlled trial. Medicine (Baltimore). 2016 Aug;95(35):e4743. doi: 10.1097/MD.0000000000004743. PMID 27583920
- [Background] Cherian MN, Mathews MP, Chandy MJ. Local wound infiltration with bupivacaine in lumbar laminectomy. Surg Neurol. 1997 Feb;47(2):120-2; discussion 122-3. doi: 10.1016/s0090-3019(96)00255-8. PMID 9040811
- [Background] Hernandez-Palazon J, Tortosa Serrano JA, Burguillos Lopez S, Molero Molero E. [Infiltration of the surgical wound with local anesthetic for postoperative analgesia in patients operated on for lumbar disc herniation. Comparative study of ropivacaine and bupivacaine]. Rev Esp Anestesiol Reanim. 2001 Jan;48(1):17-20. Spanish. PMID 11234601
- [Background] Gurbet A, Bekar A, Bilgin H, Korfali G, Yilmazlar S, Tercan M. Pre-emptive infiltration of levobupivacaine is superior to at-closure administration in lumbar laminectomy patients. Eur Spine J. 2008 Sep;17(9):1237-41. doi: 10.1007/s00586-008-0676-z. Epub 2008 Apr 19. PMID 18425538
- [Background] Ozyilmaz K, Ayoglu H, Okyay RD, Yurtlu S, Koksal B, Hanci V, Erdogan G, Turan IO. Postoperative analgesic effects of wound infiltration with tramadol and levobupivacaine in lumbar disk surgeries. J Neurosurg Anesthesiol. 2012 Oct;24(4):331-5. doi: 10.1097/ANA.0b013e3182611a1d. PMID 22759866
- [Background] Chae SU, Kim TK, Shim DM, Kim YJ, Choi DH. Is complex regional pain syndrome a cause of post-operative syndrome in the lumbar spine? - a case report -. Asian Spine J. 2009 Dec;3(2):101-5. doi: 10.4184/asj.2009.3.2.101. Epub 2009 Dec 31. PMID 20404955
- [Background] Yalbuzdag SA, Erol AM, Sengul I, Celik C, Solum S, Adilay HU, Gungor B. Temperament and Character Profile in Failed Back Surgery Syndrome: A Cross-Sectional Clinical Study. Turk Neurosurg. 2016;26(6):912-917. doi: 10.5137/1019-5149.JTN.13679-14.0. PMID 27476913
- [Result] Gruenewald M, Herz J, Schoenherr T, Thee C, Steinfath M, Bein B. Measurement of the nociceptive balance by Analgesia Nociception Index and Surgical Pleth Index during sevoflurane-remifentanil anesthesia. Minerva Anestesiol. 2015 May;81(5):480-9. Epub 2014 Jul 17. PMID 25032676